CLINICAL TRIAL: NCT01734239
Title: A Phase III, Open-Label Clinical Trial to Study the Safety and Immunogenicity of V110 in Subjects 50 Years of Age and Older and in Subjects 2 to 49 Years of Age at Increased Risk for Pneumococcal Disease, From the Russian Population
Brief Title: A Phase III Clinical Trial to Study the Safety and Immunogenicity of Pneumovax™ 23 (V110) in Participants From the Russian Population (V110-018)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V110-018
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 2,4,5,4'-tetrachlorodiphenylsulfoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pneumovax™ 23: Participants Between 2 and 49 Years (Experimental): Participants received a single, 0.5-mL intramuscular injection of Pneumovax™ 23 on Day 1
  Interventions: Biological: Pneumovax™ 23
- Pneumovax™ 23: Participants >=50 Years (Experimental): Participants received a single, 0.5-mL intramuscular injection of Pneumovax™ 23 on Day 1
  Interventions: Biological: Pneumovax™ 23

INTERVENTIONS:
Biological: Pneumovax™ 23 — Vaccine contains 25 µg of each of the 23 pneumococcal polysaccharides serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19F, 19A, 20, 22F, 23F, and 33F
  Other Names: V110

SUMMARY:
The purpose of this study is to determine if Pneumovax™ 23 (V110) is safe and immunogenic in participants from the Russian population who are 50 years of age and older or 2 to 49 years of age and at increased risk for pneumococcal disease

ELIGIBILITY:
Inclusion Criteria:

* For participants 50 years of age or older: any underlying chronic illness must be in stable condition
* For participants 2 to 49 years of age: participant has an increased risk for pneumococcal disease as a result of one of the following: chronic cardiovascular disease, chronic pulmonary disease, diabetes mellitus, alcoholism, chronic liver disease, cerebrospinal fluid leaks, functional or anatomic asplenia, sickle cell anemia, living in a special environment or social setting such as crowded, closed communities
* Male, or female not of reproductive potential, or female of reproductive potential who agrees to remain abstinent or to use 2 acceptable methods of contraception through 6 weeks after study vaccination

Exclusion Criteria:

* Received prior vaccination with pneumococcal vaccine
* Has known or suspected immune dysfunction or conditions associated with immunosuppression, or is receiving immunosuppressive chemotherapy, including long-term systemic corticosteroids
* Has history of autoimmune disease
* Received a licensed live virus vaccine within 3 months before or is scheduled within 3 months after study vaccination
* Received a licensed inactivated vaccine within 28 days before or is scheduled within 28 days after study vaccination
* Received an investigational drug or other investigational vaccine within 2 months before or is scheduled within 28 days after study vaccination (3 months if a live virus vaccine)
* Received any blood product or immunoglobulin preparation within 6 months before or 28 days after study vaccination
* Hospitalized for acute illness within 3 months before study vaccination
* Is a pregnant woman or nursing mother
* History of invasive pneumococcal disease or of other culture-positive pneumococcal disease
* History of fever illness within 3 days before study vaccination
* Received antibiotic therapy for any acute illness within 7 days before study vaccination
* Hypersensitivity to any components of the vaccine, including phenol

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2013-10-22 (Actual); Study Completion 2013-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ciprero K, Zykov KA, Briko NI, Shekar T, Sterling TM, Bitieva E, Stek JE, Musey L. Safety and immunogenicity of a single dose 23-valent pneumococcal polysaccharide vaccine in Russian subjects. Hum Vaccin Immunother. 2016 Aug 2;12(8):2142-2147. doi: 10.1080/21645515.2016.1165373. Epub 2016 May 5. PMID 27149114
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V110-018&kw=V110-018&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Pneumovax™ 23: Participants Between 2 and 49 Years; Pneumovax™ 23: Participants >=50 Years: Participants received a single 0.5 mL intramuscular injection on Day 1
Period: Overall Study
Arm/Group | Pneumovax™ 23: Participants Between 2 and 49 Years | Pneumovax™ 23: Participants >=50 Years
Started | 52 | 50
Completed | 52 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pneumovax™ 23: Participants Between 2 and 49 Years | Pneumovax™ 23: Participants >=50 Years | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.2 (15.3) | 60.4 (7.7) | 40.4 (23.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 36 | 29 | 65

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration of Antibodies to Pneumococcal Serotypes Contained in the Vaccine
Description: Serum antibodies to pneumococcal serotypes were measured by enzyme-linked immunosorbent assays
Time Frame: Prevaccination and Day 28 after vaccination
Population: The per protocol immunogenicity population included all enrolled participants except 2 who were excluded because blood samples were collected outside the allowable day range
Measure: Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Pneumovax™ 23: Participants Between 2 and 49 Years | Pneumovax™ 23: Participants >=50 Years
Number analyzed (Participants) | 52 | 48
ug/mL
  Serotype 1 prevaccination | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.3]
  Serotype 1 Day 28 postvaccination | 4.1 [3.0 to 5.4] | 2.5 [1.7 to 3.8]
  Serotype 6B prevaccination | 0.5 [0.4 to 0.8] | 0.6 [0.5 to 0.8]
  Serotype 6B Day 28 postvaccination | 2.7 [1.8 to 3.9] | 5.3 [3.4 to 8.5]
  Serotype 14 prevaccination | 1.3 [0.8 to 2.0] | 3.6 [2.5 to 5.1]
  Serotype 14 Day 28 postvaccination | 13.2 [8.7 to 20.1] | 32.7 [22.7 to 47.3]
  Serotype 19F prevaccination | 1.5 [1.1 to 2.2] | 1.5 [1.1 to 2.1]
  Serotype 19F Day 28 postvaccination | 12.6 [9.0 to 17.8] | 9.9 [7.0 to 14.1]
  Serotype 23F prevaccination | 0.6 [0.4 to 1.0] | 1.1 [0.7 to 1.5]
  Serotype 23F Day 28 postvaccination | 5.3 [3.6 to 7.7] | 8.1 [5.3 to 12.4]

2. Primary Outcome: Percentage of Participants With >=2-fold Increase From Prevaccination to Postvaccination in Antibodies to Pneumococcal Serotypes Contained in the Vaccine
Description: Serum antibodies to pneumococcal serotypes were measured by enzyme-linked immunosorbent assays. A >=2-fold increase in serum antibody is a marker for serologic response to pneumococcal vaccination in adults.
Time Frame: Day 28 postvaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pneumovax™ 23: Participants Between 2 and 49 Years | Pneumovax™ 23: Participants >=50 Years
Number analyzed (Participants) | 52 | 48
Percentage of participants
  Serotype 1 | 96.2 [86.8 to 99.5] | 87.5 [74.8 to 95.3]
  Serotype 6B | 76.9 [63.2 to 87.5] | 89.6 [77.3 to 96.5]
  Serotype 14 | 88.5 [76.6 to 95.6] | 89.6 [77.3 to 96.5]
  Serotype 19F | 82.7 [69.7 to 91.8] | 79.2 [65.0 to 89.5]
  Serotype 23F | 80.8 [67.5 to 90.4] | 87.5 [74.8 to 95.3]

3. Primary Outcome: Number of Participants With Elevated Body Temperature (>=37.6 °C Axillary / >=38.0 °C Oral or Equivalent)
Time Frame: Up to 5 days postvaccination
Population: The All Subjects as Treated population included all enrolled participants
Measure: Number; unit: Number of participants
Arm/Group | Pneumovax™ 23: Participants Between 2 and 49 Years | Pneumovax™ 23: Participants >=50 Years
Number analyzed (Participants) | 52 | 50
Number of participants | 1 | 0

4. Primary Outcome: Number of Participants Reporting an Injection-site or Systemic Adverse Experience That Was Reported by >=4 Participants
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the sponsor's product, is also an AE. Injection-site or systemic AEs that occurred in >=4 participants were reported for this endpoint.
Time Frame: Up to Day 14 postvaccination
Population: The All Subjects as Treated population included all enrolled participants
Measure: Number; unit: Number of participants
Arm/Group | Pneumovax™ 23: Participants Between 2 and 49 Years | Pneumovax™ 23: Participants >=50 Years
Number analyzed (Participants) | 52 | 50
Number of participants | 16 | 5

5. Primary Outcome: Number of Participants Reporting Serious Adverse Experiences
Description: A serious AE (SAE) is an AE that 1) results in death, 2) is life threatening, 3) results in a persistent or significant disability or incapacity, 4) results in or prolongs an existing inpatient hospitalization, 5) is a congenital anomaly or birth defect, 6) is a cancer, 7) is an overdose, or 8) is another important medical event which, based on appropriate medical judgment, may jeopardize the participant and may require medical or surgical intervention
Time Frame: Up to Day 28 postvaccination
Population: The All Subjects as Treated population included all enrolled participants
Measure: Number; unit: Number of participants
Arm/Group | Pneumovax™ 23: Participants Between 2 and 49 Years | Pneumovax™ 23: Participants >=50 Years
Number analyzed (Participants) | 52 | 50
Number of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse experiences were collected through Day 14 postvaccination; serious adverse experiences were collected through Day 28 postvaccination
Groups:
- Pneumovax™ 23: Participants received a single 0.5 mL intramuscular injection on Day 1
Arm/Group | Pneumovax™ 23
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 14/102
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumovax™ 23 (N=102)
Injection site pain (General disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.